CLINICAL TRIAL: NCT00001054
Title: A Phase I Trial to Evaluate the Pharmacokinetics, Safety, and Tolerance of Valacyclovir HCl in HIV-1 Infected Children With Herpes Simplex Infections or Varicella/Zoster Infections
Brief Title: The Safety and Effectiveness of Valacyclovir HCl in the Treatment of Herpes Simplex or Varicella/Zoster Infections in HIV-1 Infected Children
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 253; 11230 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Herpes Simplex; HIV Infections; Chickenpox
Keywords: Herpes Zoster; AIDS-Related Opportunistic Infections; Herpes Simplex; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; valacyclovir; Chickenpox
MeSH Terms: conditions — Herpes Simplex; HIV Infections; Chickenpox; Herpes Zoster; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Valacyclovir

INTERVENTIONS:
Drug: Valacyclovir hydrochloride

SUMMARY:
To obtain tolerance, safety, and pharmacokinetic data for oral valacyclovir hydrochloride ( 256U87 ) in HIV-1 infected children with herpes simplex virus infections ( cold sores ) and/or varicella / zoster virus infections ( chicken pox / shingles ).

Varicella and zoster are common problems in HIV-infected children. It is believed that chronic oral therapy with acyclovir may result in subtherapeutic concentrations of acyclovir, resulting in resistance to that drug. Valacyclovir hydrochloride, which converts to acyclovir in the body, increases acyclovir bioavailability by 3-5 fold.

DETAILED DESCRIPTION:
Varicella and zoster are common problems in HIV-infected children. It is believed that chronic oral therapy with acyclovir may result in subtherapeutic concentrations of acyclovir, resulting in resistance to that drug. Valacyclovir hydrochloride, which converts to acyclovir in the body, increases acyclovir bioavailability by 3-5 fold.

In the first cohort, patients with stable herpes simplex virus receive valacyclovir hydrochloride at 1 of 2 doses, depending on body surface area (BSA), for 10 days. If acceptable safety is seen at this dose level, a second cohort of patients with stable herpes simplex virus receive a higher dose, depending on BSA, for 10 days. A third cohort of patients with varicella or zoster receive a selected dose based on results from the previous cohorts.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiretrovirals.
* PCP prophylaxis.
* IVIG, G-CSF, and erythropoietin.

Concurrent Treatment:

Allowed:

* Transfusions.

Patients must have:

* Localized mucocutaneous herpes simplex OR undisseminated varicella or zoster.
* HIV positive. NOTE: Varicella patients must NOT have AIDS.
* CD4 count >= 100 cells/mm3 (herpes simplex or zoster patients) OR >= 250 cells/mm3 (varicella patients).
* BSA > 0.6 m2.
* Ability to swallow solid dosage formulations.

Prior Medication:

Allowed:

* Prior VZV immune globulin and/or IVIG.
* Antiretrovirals if at a stable dose for at least 14 days.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Clinical evidence of pneumonitis.
* Severe abdominal pain or back pain.
* Encephalopathy.
* Hemorrhagic varicella.
* Zoster involving ophthalmic branch of trigeminal nerve.
* Severe gastrointestinal disorder.

Concurrent Medication:

Excluded:

* Agents with potential activity against HSV or VZV, such as acyclovir, famciclovir, ganciclovir, foscarnet, and sorivudine.
* Probenecid.
* Aspartamine within 48 hours prior to pharmacokinetic samplings.

Patients with the following prior conditions are excluded:

* Grade 2 creatinine value within the past 30 days.
* Grade 3 hematologic or hepatic values within the past 30 days.
* Prior hypersensitivity and/or allergic reaction to acyclovir.
* Grade 3 or 4 mental status changes within the past 30 days.

Prior Medication:

Excluded:

* Acyclovir within 1 week prior to study entry.
* Steroids within 4 weeks prior to onset of varicella lesions.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Study Completion 2001-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keller MA, Study Chair; Bryson Y, Study Chair; Gershon A, Study Chair

REFERENCES:
- [Background] von Seidlein L, Gillette SG, Bryson Y, Frederick T, Mascola L, Church J, Brunell P, Kovacs A, Deveikis A, Keller M. Frequent recurrence and persistence of varicella-zoster virus infections in children infected with human immunodeficiency virus type 1. J Pediatr. 1996 Jan;128(1):52-7. doi: 10.1016/s0022-3476(96)70427-4. PMID 8551421
- [Background] Cohen JI, Brunell PA, Straus SE, Krause PR. Recent advances in varicella-zoster virus infection. Ann Intern Med. 1999 Jun 1;130(11):922-32. doi: 10.7326/0003-4819-130-11-199906010-00017. PMID 10375341